CLINICAL TRIAL: NCT01152255
Title: A Multiple Dose Clinical Trial to Study the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MK6186 in HIV-1 Infected Patients
Brief Title: MK6186 in HIV-1 Infected Patients (MK-6186-007 AM2)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6186-007; 2010_542; 2010-020829-41 (EudraCT Number)
Record Dates: First submitted 2010-06-25; First posted 2010-06-29 (Estimated); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: HIV-1 Infection
Keywords: Treatment of HIV-1 Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Panel A - MK6186 40 mg (Experimental): MK6186 40 mg
  Interventions: Drug: MK6186
- Panel A - Placebo (Placebo Comparator): placebo
  Interventions: Drug: Comparator: Placebo
- Panel B - MK6186 150 mg (Experimental): MK6186 150 mg
  Interventions: Drug: MK6186
- Panel B - Placebo (Placebo Comparator): placebo
  Interventions: Drug: Comparator: Placebo
- Panel C - MK6186 <=150 mg (Experimental): MK6186 <=150 mg
  Interventions: Drug: MK6186
- Panel C - Placebo (Placebo Comparator): placebo
  Interventions: Drug: Comparator: Placebo
- Panel D - MK6186 <=150 mg (Experimental): MK6186 <=150 mg
  Interventions: Drug: MK6186
- Panel D - Placebo (Placebo Comparator): placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: MK6186 — Panel A: 40 mg oral dose once daily for 7 days Panel B: 150 mg oral dose once daily for 7 days Panel C: Oral Dose <= 150 mg once daily for 7 days (dose level will be determined based on pharmacokinetic and pharmacodynamic results of panel A and B) Panel D: Oral Dose <= 150 mg once twice or three times daily for 7 days (dose level and dose frequency will be determined based on pharmacokinetic and pharmacodynamic results of panel A, B and C)
  Arms: Panel A - MK6186 40 mg; Panel B - MK6186 150 mg; Panel C - MK6186 <=150 mg; Panel D - MK6186 <=150 mg
Drug: Comparator: Placebo — Placebo tablets taken orally for seven day
  Arms: Panel A - Placebo; Panel B - Placebo; Panel C - Placebo; Panel D - Placebo

SUMMARY:
This study will evaluate the safety and tolerability of MK6186 and the change from baseline in plasma HIV-1 RNA after seven consecutive days of dosing.

ELIGIBILITY:
Inclusion Criteria:

* Other than HIV infection, patient's baseline health is judged to be stable
* Patient is documented HIV-1 positive
* Patient has not received an investigational agent or licensed ART with in the past 30 days

Exclusion Criteria:

* Patient has a history of stroke, chronic seizures, or major neurological disease
* Patient has a history of cancer
* Patient has used any immune therapy agents or immunosuppressive therapy within the past month
* Patient requires or anticipates the use of any prescription or non-prescription drugs during the study
* Patient has a current diagnosis of acute hepatitis, has a history of Hepatitis C or has positive Hepatitis B surface antigen
* Patient consumes excessive amounts of alcohol (greater than 3 servings per day) or caffeine (greater than 6 servings per day)
* Patient is an excessive smoker (more than 10 cigarettes per day)
* Patient has had major surgery, donated blood or participated in another investigational study within the past 4 weeks

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-10-10 (Actual); Primary Completion 2011-06-30 (Actual); Study Completion 2011-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in plasma HIV-1 RNA | Baseline and Day 7
Safety and tolerability of MK6186 measured by number of clinical and laboratory adverse experiences | through Day 21

SECONDARY OUTCOMES:
C(24 hour) of MK6186 | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Schurmann D, Huser A, Pfafflin F, Cilissen C, De Lepeleire I, Larson PJ, Anderson MS, Rizk ML, Hofmann J, Daumer M, Stegemann MS, Stoch SA, Wagner F, Iwamoto M. A Randomized, Double-Blind, Placebo-Controlled, Short-Term Monotherapy Study of MK-6186, an HIV-1 Non-Nucleoside Reverse Transcriptase Inhibitor, in Treatment-Naive HIV-Infected Participants. AIDS Res Hum Retroviruses. 2025 Jan;41(1):11-19. doi: 10.1089/AID.2023.0152. Epub 2024 Oct 3. PMID 39291814